CLINICAL TRIAL: NCT01512316
Title: The Effect of D-cycloserine on Fear Learning and Extinction
Brief Title: Exploring Learning and Unlearning of Fear
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was cancelled
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IMDCSACQEXT
Record Dates: First submitted 2011-12-22; First posted 2012-01-19 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2016-05

CONDITIONS: Healthy Individuals
Keywords: Fear; Cycloserine; Conditioning; Functional neuroimaging; Anxiety disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Cycloserine; Lactose; Functional Neuroimaging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- d-Cycloserine Acquisition (Active Comparator): d-Cycloserine will be given on day1, before acquisition
  Interventions: Drug: d-Cycloserine; Genetic: Saliva sample; Other: Functional neuroimaging (fMRI)
- d-Cycloserine Extinction (Active Comparator): d-Cycloserine will be administered on day2, before extinction
  Interventions: Drug: d-Cycloserine; Genetic: Saliva sample; Other: Functional neuroimaging (fMRI)
- Placebo (Placebo Comparator): A placebo pill will be administered on day1 and 2
  Interventions: Drug: Lactose pill; Genetic: Saliva sample; Other: Functional neuroimaging (fMRI)

INTERVENTIONS:
Drug: d-Cycloserine — 250mg, one dose, 2hrs prior to fMRI
  Other Names: Cycloserine, King Pharmaceuticals Ltd
  Arms: d-Cycloserine Acquisition; d-Cycloserine Extinction
Drug: Lactose pill — one dose, 2hrs prior to fmri
  Arms: Placebo
Genetic: Saliva sample — Buccal cell material will be sampled from all participants on day3
  Other Names: Whatman's Sterile Omni Swabs (www.whatman.com)
Other: Functional neuroimaging (fMRI)

SUMMARY:
The present study investigates the effect of d-cycloserine on learning and unlearning of fear in healthy humans and its underlying effect on the amygdala.

As a second objective, the effect of genotype on fear learning will be studied.

DETAILED DESCRIPTION:
A growing body of evidence suggests that the extinction of fear is mediated by the N-methyl-D-aspartate (NMDA) receptor activity in the basolateral amygdala. Intra-amygdala infusions of antagonists of this glutamate receptor in small animals (eg: rats, mice) have demonstrated a blockage of fear acquisition and extinction. Agonists, on the other hand, facilitate conditioned fear extinction.

The animal studies are all based on the simple fear learning paradigm of conditioning. However, it is not clear that human anxiety disorders are based on prior conditioning encounter. Therefore it is important to disentangle the effect of DCS on acquisition and extinction in the context of a simple learning paradigm, particular its effect on the human amygdala.

ELIGIBILITY:
Inclusion Criteria:

* No axis I diagnosis compatible with the DSM-IV by means of a structured diagnostic interview
* Right-handed

Exclusion Criteria:

* Current psychopharmacological or psychological treatment.
* The presence of a physical/medical condition that may interfere with the study.
* A contraindication for the use of DCS
* Pacemaker, medication pump (such as insulin pump), hearing aid, removable prosthodontics
* Metal in or on body (such as acupuncture needles, artificial limbs, stents, metal splints, clips, implanted electrodes, tattoos, or piercings)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
change in BOLD-signal during a fear conditioning task | t0, t+24, t+48
  Subjects will participate in a 3-day experiment. Day1 (t0): Acquisition Day2 (T+24): extinction Day3 (T+48): re-exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University Leuven, Departement of Radiology, Leuven, Belgium